CLINICAL TRIAL: NCT02244567
Title: Effect of Metformin Therapy on Serum Under-carboxylated Osteocalcin in Hyperandrogenic Lean PCOS Women
Brief Title: Effect of Metformin Therapy on Serum Under-carboxylated Osteocalcin Levels in Hyperandrogenic Lean Polycystic Ovarian Syndrome Women
Acronym: U-C OC IN PCOS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Lecturer of Obstetrics and Gynecology, Beni-Suef University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Beni-Suef 4
Record Dates: First submitted 2014-09-13; First posted 2014-09-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Pharmaceutical Preparations; Vitamins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metformin (Active Comparator): Cidophage 850 mg twice daily for three months will be given to the patientwith PCOS.
  Interventions: Drug: Metformin 850 mg twice daily for 3 months
- Serum under-carboxylated osteocalcin (Active Comparator): Serum uc-oc will be measured before and after 3 months of treatment with cidophage.
  Interventions: Procedure: Serum uc-oc
- Placebo (Active Comparator): Other group of patients with high serum UC-OC will be given a placebo.
  Interventions: Other: drug

INTERVENTIONS:
Drug: Metformin 850 mg twice daily for 3 months — This drug is insulin sensitizing agent which will be given twice daily orally for 3 months for PCOS patients.
  Other Names: Cidophage
  Arms: Metformin
Procedure: Serum uc-oc — Serum uc-oc is a bone biomarker involved in incraesing insulin in pathophysiology of PCOS. It will be measured in serum of pcos patients before and after treatment with metformin for 3 months.
  Other Names: Serum undercarboxylated-osteocalcin
  Arms: Serum under-carboxylated osteocalcin
Other: drug — This group of patients will receive any type of vitamin as a placebo to compare with effect of Metformin on serum UC-OC.
  Other Names: vitamin
  Arms: Placebo

SUMMARY:
High ucOC may favor insulin release in lean hyperandrogenic women to compensate for impaired insulin sensitivity. Meformin is an insulin sensitizing agent will be given for these women trying to interfere with the pathophysiology of PCOS in these women as followed up by serum UC-OC levels.

DETAILED DESCRIPTION:
Under-carboxylated osteocalcin (ucOC), the precursor substrate of bone biomarker OC is a potent regulator of energy metabolism by promoting insulin production and adiponectin synthesis and decreasing fat stores.UcOC has a potential role in the physiopathology of polycystic ovary syndrome (PCOS), a common disorder defined by the constellation of anovulation, insulinresistance, hyperinsulinemia, obesity and androgen excess.Circulating ucOC concentration is related to key endocrine PCOS characteristics in a weight-dependent manner. Within the bone-pancreas loop, high ucOC may favor insulin release in lean hyperandrogenic women to compensate for impaired insulin sensitivity.We will investigate serum uc-OC responses to insulin sensitizing therapies in lean hyperandrogenic polycystic ovary syndrome (PCOS).

ELIGIBILITY:
Inclusion Criteria:

* Lean women BMI 25 or less
* Hyperandrogenic clinically and/or biochemically.
* Androgen Excess-Polycystic Ovary Syndrome (AE-PCOS) Society 2006 criteria

Exclusion Criteria:

* BMI more than 20
* Other causes of hyperandrogenism
* Other causes of metabolic disorders or diabetes.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
High Serum under-carboxylated osteocalcin | 3 months
  Hyperandrogenic lean women will be diagnosed as PCOS according to Androgen Excess-Polycystic Ovary Syndrome (AE-PCOS) Society 2006 criteria.Serum uc-oc will be assayed when it is found to be high, metformin therapy for three months will be given to these women. Serum uc-oc will be measured again and effect of therapy will be interpreted.

SECONDARY OUTCOMES:
Metformin therapy | 3 months
  Cidophage 850 mg twice daily will be given for three months to pcos patients who are hyperandrogenic and lean then serum uc-oc will be measured after therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Nesreen Abdel Fattah Abdullah Shehata, Cairo, Egypt

REFERENCES:
- See also: Pepene CE. Serum under-carboxylated osteocalcin levels in women with polycystic ovary syndrome: weight-dependent relationships with endocrine and metabolic traits. J Ovarian Res. 2013;6(1):4. — http://www.ncbi.nlm.nih.gov/